CLINICAL TRIAL: NCT03450161
Title: Hyperalgesia, Persistent Pain, and Fentanyl Dosing in On-Pump Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGO/2017/005; 2017-003278-15 (EudraCT Number)
Record Dates: First submitted 2018-01-29; First posted 2018-03-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hyperalgesia; Opioid Use; Pain, Postoperative; Pain, Chronic
MeSH Terms: conditions — Hyperalgesia; Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, three arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only an otherwise uninvolved anesthesiologist will know dosing schemes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-Dose Bolus of Fentanyl (Experimental): 5 minutes prior to sternotomy, patients will receive a fentanyl bolus of 20 mcg/kg BW (verum) and a perfusion pump with sodium chloride (NaCl 0.9%; placebo) will be begun according to the Shibutani dosing scheme.
  As in the other arms, patients will be induced with 3mcg/kg BW fentanyl and the treating physician may administer boli on an "as needed" basis.
  Interventions: Drug: Fentanyl dosing schemes
- Low-Dose Bolus of Fentanyl (Experimental): 5 minutes prior to sternotomy, patients will receive a fentanyl bolus of 3 mcg/kg BW (verum) and a perfusion pump with sodium chloride (NaCl 0.9%; placebo) will be begun according to the Shibutani dosing scheme.
  As in the other arms, patients will be induced with 3mcg/kg BW fentanyl and the treating physician may administer boli on an "as needed" basis.
  Interventions: Drug: Fentanyl dosing schemes
- Continuous Dose of Fentanyl (Experimental): 5 minutes prior to sternotomy, patients will receive a NaCl 0.9% bolus (placebo) and a perfusion pump with fentanyl (verum) will be begun according to the Shibutani dosing scheme.
  As in the other arms, patients will be induced with 3mcg/kg BW fentanyl and the treating physician may administer boli on an "as needed" basis.
  Interventions: Drug: Fentanyl dosing schemes

INTERVENTIONS:
Drug: Fentanyl dosing schemes — We routinely use fentanyl as the opioid of choice in CABG surgery. However, how much and whether or not to apply it in boli or continuously remain uncertain. We will apply 3 routinely used fentanyl dosing schemes in our hospital. To blind care-givers and patients, in each of the arms a bolus and a continous injection will occur, as delineated in the treatment arms.

SUMMARY:
Randomized, double-blinded, three arm study in adult patients undergoing first time coronary artery bypass grafting (CABG) surgery with median sternotomy. The investigators will examine the effects of three fentanyl dosing schemes (high-dose bolus, low-dose bolus, continuous dose) on the area of hyperalgesia and allodynia at 24 and 48h as well as on persisting pain at 3, 6, and 12 months. Additionally, the investigators will measure fentanyl concentrations throughout anesthesia.

DETAILED DESCRIPTION:
A prospective, randomized, double-blinded (patient, anesthesiologist, assessor) clinical study. This study will examine three different clinically used application schemes of fentanyl, an opioid used as the standard of care in routine practice. Patients will be randomized to receive one of the following three treatment arms for anesthesia maintenance (pre-sternotomy):

1. High-dose fentanyl bolus (20 µg/kg of body weight [BW]; e.g. 70kg 1400 µg or 1.4mg)
2. Low-dose fentanyl bolus (3 µg/kg BW; e.g. 70kg 210 µg or 0.2mg)
3. Continuous fentanyl application by Shibutani scheme

   This study will include data from 69 adult patients (23 per arm) undergoing first time, elective, on-pump CABG surgery with median sternotomy and central cannulation.

   Following randomization by the sealed envelope technique, fentanyl kits will be drawn up by an anesthesiologist not involved in patient care or outcome assessment. Patients with preexisting chronic pain, opioids in the last 30 days, a BMI>36kg/m2, sleep apnoea, renal failure (clearance <30ml/min), with neuraxial anesthesia, pregnant, with planned wound infiltration, known allergies/intolerance to opioids, and unable to understand pin-prick testing will be excluded.

   At induction, all patients will receive a standard 3 µg/kg bolus of fentanyl (not study medication, but rather standard of care). 5 minutes prior to sternotomy, the patient will receive analgesia maintenance (one of the three fentanyl study arms). Clinicians will at all times be able to administer a bolus of fentanyl on a perceived "as needed" basis (not study medication, but rather standard of care).

   The primary objective of this trial is to assess whether or not different intraoperative dosing schemes of fentanyl during on-pump CABG surgery influence the area of hyperalgesia as measured by sternal pin-prick testing on the first postoperative day. As the mechanisms causing opioid-induced analgesia are poorly understood but appear to be dosis-related, the investigators will examine 3 clinically used fentanyl application schemes in cardiac surgery: 1) a high-dose bolus group, 2) a low-dose bolus group, and 3) a low-dose continuous infusion group.

   [i.e. does fentanyl dosing influence the area of hyperalgesia?]

   The secondary objectives of this trial are 1) to explore the intraoperative concentrations of fentanyl in these various dosing schemes during and after extracorporeal circulation (ECC).

   [i.e. determine the time course of fentanyl with ECC and its association with hyperalgesia; explorative] 2) to explore a possible association between fentanyl dosing, hyperalgesia, and persisting pain 3, 6, and 12 months after surgery.

   [i.e. clinical implication on persistent/chronic pain; explorative]

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients aged ≥18 years
* Undergoing first-time, elective, on-pump CABG surgery with median sternotomy and central cannulation.

Exclusion Criteria:

* Documentation of preexisting chronic pain as per electronic record
* Use of opioids in the last 30 days or history/documentation of opioid abuse as per electronic record
* BMI > 35kg/m2 or history of obstructive sleep apnea syndrome
* Patients with renal failure (clearance < 30 ml/min)
* Neuraxial anesthesia
* Pregnancy
* Planned wound infiltration with local anesthetics
* Known drug allergies or intolerance to fentanyl or other opioids
* Expected to be unable to understand pinprick/allodynia testing / follow-up questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Area of hyperalgesia at 24h | 24 hours after surgery (+/- 3 hours)
  Determination of secondary, wound hyperalgesia by pin prick (256mN von Frey filament)

SECONDARY OUTCOMES:
Area of hyperalgesia at 48h | 48 hours after surgery (+/- 3 hours)
  Determination of secondary, wound hyperalgesia by pin prick (256mN von Frey filament)
Area of allodynia at 24h | 24 hours after surgery (+/- 3 hours)
  Determination of allodynia by cotton swab
Area of allodynia at 48h | 48 hours after surgery (+/- 3 hours)
  Determination of allodynia by cotton swab
Persistent Pain at 3 months | 3 months after surgery (+/- 1 week)
  Validated questionnaire to assess pain after by1) mail and 2) phone follow-up
Persistent Pain at 6 months | 6 months after surgery (+/- 1 week)
  Validated questionnaire to assess pain after by1) mail and 2) phone follow-up
Persistent Pain at 12 months | 12 months after surgery (+/- 1 week)
  Validated questionnaire to assess pain after by1) mail and 2) phone follow-up
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 5 min. (+/- 1 min) prior to sternotomy, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run as specified by the time frame of this outcome and the following outcomes.
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 5 min. (+/- 1 min) after fentanyl/placebo bolus, given just prior to sternotomy
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 30 min. (+/- 1 min) after fentanyl/placebo bolus, given just prior to sternotomy
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | just prior (<1min) to start of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 5 min. (+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 20 min. (+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 40 min.(+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 60 min.(+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 80 min. (+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 100 min. (+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 120 min.(+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 140 min.(+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 160 min.(+/- 1 min) after begin of pump run, a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | 5 min.(+/- 1 min) after end of pump run,a surgical step
  Fentanyl will be measured from samples taken prior to, during, and after a pump run
Description of perioperative fentanyl concentrations with on-pump extra corporeal circulation | end of surgery (+/- 5 min)
  Fentanyl will be measured from samples taken prior to, during, and after a pump run

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided